CLINICAL TRIAL: NCT00642486
Title: Portable Monitoring in the Diagnosis and Management of Obstructive Sleep Apnea
Brief Title: Portable Monitoring for Diagnosis and Management of Sleep Apnea
Acronym: HomePAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: University Hospitals Cleveland Medical Center (Other); The Cleveland Clinic (Other); MetroHealth Medical Center (Other); University of Washington (Other); University of Minnesota (Other); Northwestern University (Other); University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASMF 38-PM-07
Record Dates: First submitted 2008-03-24; First posted 2008-03-25 (Estimated); Last update posted 2025-08-05 (Actual); Status verified 2008-03

CONDITIONS: Sleep Apnea, Obstructive
Keywords: treatment; positive airway pressure; compliance; cost effectiveness; clinical trial
MeSH Terms: conditions — Sleep Apnea, Obstructive; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): laboratory-based testing
  Interventions: Other: Standard polysomnography (PSG)
- 2 (Active Comparator): home-based testing
  Interventions: Other: Portable (Embla Embletta X30 system and Respironic REMStar Auto M series with CFlex)

INTERVENTIONS:
Other: Portable (Embla Embletta X30 system and Respironic REMStar Auto M series with CFlex) — portable, home-based using the Embla Embletta X30 system as the diagnostic device and the Respironic REMStar Auto M series with CFlex as the PAP titration device.
  Arms: 2
Other: Standard polysomnography (PSG) — laboratory-based testing
  Arms: 1

SUMMARY:
This multi-site project compares compares the efficiency of a home-based portable monitoring strategy to a standard of care sleep laboratory-based strategy for the diagnosis and positive airway pressure treatment of obstructive sleep apnea in adults.

DETAILED DESCRIPTION:
The study is a randomized, parallel group, unblinded, multicenter study that compares two approaches [home-based, portable monitoring (PM) versus attended, laboratory-based polysomnography (PSG) (Lab)] in adults, at least 18 years of age, with a moderate to high probability of obstructive sleep apnea (OSA) and who have been referred to sleep medicine specialists at AASM-accredited sleep centers for evaluation and/or management. The study is designed to compare the utility of the two approaches (PM group vs. Lab group) for the diagnosis and management of OSA in adults. Approximately 372 eligible adults will be randomized at screening to either the PM or Lab arm (186 per arm), undergo baseline OSA testing to confirm diagnosis and study eligibility, then receive positive airway pressure (PAP) titration studies to determine the level of pressure needed to treat their OSA. For qualifying participants, the titration study will be lab-based in the Lab group and be home-based using a commercially available portable, automatic PAP device (APAP) in the PM group. All qualifying study participants will have access to study CPAP equipment and supplies to treat their OSA. Primary outcomes (time from diagnosis to effective treatment, patient outcomes, and relative resource utilization) are determined at 1 and 3 months after starting CPAP treatment. Study participants who complete all of their study visits will keep their CPAP machine at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Intermediate to high probability of having OSA based on an adjusted neck circumference > 43 cm (17 inches)
* Presence of excessive daytime sleepiness (Epworth sleepiness scale ≥ 12) Apnea-hypopnea index >= 15 on diagnostic testing to continue in study

Exclusion Criteria:

* Severe chronic insomnia, other condition with < 4 hrs of sleep per night
* Unstable medical conditions
* Major psychiatric diagnosis
* Unable to undergo home testing
* Concerns about unsafe driving
* Severe COPD or restrictive lung disease
* Chronic narcotic use
* Alcohol abuse
* History of cataplexy
* Moderate to severe restless legs syndrome symptoms
* Pre-existing diagnosis of sleep apnea
* Prior experience with positive airway pressure treatment of sleep apnea
* Anticipated upper airway surgery or gastric bypass surgery in 4 months
* Decisional impairment for consenting
* Hypoventilation syndrome, identified in the medical record
* Waking oxygen saturation < 92%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 373 (Actual)
Dates: Start 2008-02; Primary Completion 2009-07 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Acceptance of CPAP treatment | from diagnosis to effective treatment

SECONDARY OUTCOMES:
Compliance with CPAP therapy | 1 and 3 month post acceptance

CONTACTS AND LOCATIONS:
Overall Officials: Carol L Rosen, MD, Principal Investigator — Case Western Reserve University
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Pascoe M, Bena J, Andrews ND, Auckley D, Benca R, Billings ME, Kapur VK, Iber C, Zee PC, Redline S, Rosen CL, Foldvary-Schaefer N. Dose-response relationship between positive airway pressure therapy and excessive daytime sleepiness: the HomePAP study. J Clin Sleep Med. 2022 Apr 1;18(4):1027-1034. doi: 10.5664/jcsm.9792. PMID 34870587
- [Derived] Kim RD, Kapur VK, Redline-Bruch J, Rueschman M, Auckley DH, Benca RM, Foldvary-Schafer NR, Iber C, Zee PC, Rosen CL, Redline S, Ramsey SD. An Economic Evaluation of Home Versus Laboratory-Based Diagnosis of Obstructive Sleep Apnea. Sleep. 2015 Jul 1;38(7):1027-37. doi: 10.5665/sleep.4804. PMID 26118558
- [Derived] Billings ME, Rosen CL, Auckley D, Benca R, Foldvary-Schaefer N, Iber C, Zee PC, Redline S, Kapur VK. Psychometric performance and responsiveness of the functional outcomes of sleep questionnaire and sleep apnea quality of life instrument in a randomized trial: the HomePAP study. Sleep. 2014 Dec 1;37(12):2017-24. doi: 10.5665/sleep.4262. PMID 25325491
- [Derived] Billings ME, Rosen CL, Wang R, Auckley D, Benca R, Foldvary-Schaefer N, Iber C, Zee P, Redline S, Kapur VK. Is the relationship between race and continuous positive airway pressure adherence mediated by sleep duration? Sleep. 2013 Feb 1;36(2):221-7. doi: 10.5665/sleep.2376. PMID 23372269
- [Derived] Rosen CL, Auckley D, Benca R, Foldvary-Schaefer N, Iber C, Kapur V, Rueschman M, Zee P, Redline S. A multisite randomized trial of portable sleep studies and positive airway pressure autotitration versus laboratory-based polysomnography for the diagnosis and treatment of obstructive sleep apnea: the HomePAP study. Sleep. 2012 Jun 1;35(6):757-67. doi: 10.5665/sleep.1870. PMID 22654195
- [Derived] Billings ME, Auckley D, Benca R, Foldvary-Schaefer N, Iber C, Redline S, Rosen CL, Zee P, Kapur VK. Race and residential socioeconomics as predictors of CPAP adherence. Sleep. 2011 Dec 1;34(12):1653-8. doi: 10.5665/sleep.1428. PMID 22131602